CLINICAL TRIAL: NCT05282901
Title: A Phase II, Monocentric, Single Arm Trial Evaluating the Efficacy and Safety of Pembrolizumab in Combination With Lenvatinib in Metastatic Uveal MElanoma Patients
Brief Title: Efficacy and Safety of Pembrolizumab in Combination With Lenvatinib in Metastatic Uveal MElanoma Patients (PLUME)
Acronym: PLUME
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2020-06
Record Dates: First submitted 2022-02-24; First posted 2022-03-16 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Uveal Melanoma
Keywords: Metastatic; Uveal; Melanoma; Immune; Response
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis; Melanoma | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Intervention Model Description: Monocentric, phase II trial with a single-arm of treatment in two independent cohorts with Tebentafusp-naive patients, and with patients previously treated by Tebentafusp
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metastatic Uveal MElanoma patients (Experimental): Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic uveal melanoma (UM)
  Interventions: Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution

INTERVENTIONS:
Drug: Pembrolizumab 25 MG/1 ML Intravenous Solution — Taken together, we hypothesize that combining pembrolizumab with lenvatinib in metastatic UM may target essential cellular oncogenic pathways while normalizing tumor vascularization, thus allowing an increased infiltration of the tumor by immune cells and an improved immune response.
  Other Names: Lenvatinib

SUMMARY:
Because we suspect that the benefit of anti-PD-1 in metastatic UM patients could vary according to previous exposure to Tebentafusp (better efficacy of anti-PD-1 after Tebentafusp), the combination of pembrolizumab and lenvatinib will be assessed in two independent cohorts: cohort 1 with Tebentafusp-naive patients, and cohort 2 with patients previously treated by Tebentafusp.

The study is a monocentric, phase II trial with a single-arm of treatment in each cohort.

Liver MRI and chest-abdomen-pelvis CT will be performed every 9 weeks until progressive disease (PD), followed by a Follow-up visit within 28 days after last treatment intake. Survival status will be registered after patient discontinuation.

DETAILED DESCRIPTION:
After a screening phase of up to 28 days, each participant will receive assigned study intervention of pembrolizumab (maximum of 35 cycles) plus lenvatinib until reaching a discontinuation criterion including disease progression.

Because we suspect that the benefit of anti-PD-1 in metastatic UM patients could vary according to previous exposure to Tebentafusp (better efficacy of anti-PD-1 after Tebentafusp), the combination of pembrolizumab and lenvatinib will be assessed in two independent cohorts: cohort 1 with Tebentafusp-naive patients, and cohort 2 with patients previously treated by Tebentafusp.

The study is a monocentric, phase II trial with a single-arm of treatment in each cohort.

Liver MRI and chest-abdomen-pelvis CT will be performed every 9 weeks until progressive disease (PD), followed by a Follow-up visit within 28 days after last treatment intake. Survival status will be registered after patient discontinuation.

Participants who discontinue for reasons other than radiographic PD will have post-treatment follow-up imaging for disease status until (i) PD is documented radiographically per RECIST 1.1, or (ii) a non-study anticancer treatment is initiated, or (iii) consent is withdrawn, or (iv) the participant becomes lost to follow-up.

Lenvatinib will not be stopped for complete response (CR); participants should remain on lenvatinib until the discontinuation criterion are met.

All participants will be followed for OS until death, withdrawal of consent, loss to follow-up, or the end of the study. The survival status of all the participants will be collected at the date of the Last Visit of the Last Patient.

Exploratory research on biomarkers of response or resistance will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of metastatic uveal melanoma (UM).
2. (i) Not having been treated with Tebentafusp for cohort 1 (Tebentafusp-naive patients) OR (ii) Having been previously treated with Tebentafusp for cohort 2.
3. Life expectancy > 3 months.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG has to be performed at inclusion.
5. Male participants must agree to use contraception
6. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) OR
   2. A WOCBP who agrees to follow the contraceptive guidance
7. Measurable disease based on RECIST 1.1. lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
8. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
9. Have provided a newly obtained (or archival if no systemic treatment since the sampling) core or excisional biopsy of a tumor lesion not previously irradiated.
10. Patients with French Social Security in compliance with the French law relating to biomedical research
11. All other relevant medical conditions must be well-managed and stable, in the opinion of the investigator, for at least 28 days prior to first administration of study drug.
12. Have adequate organ function as defined in the protocol.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to allocation.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, and CD137) for metastatic UM.

   In contrast, prior therapy with Tebentafusp is permitted.
3. Has recently received prior systemic anti-cancer therapy including investigational agents or biological agents [eg cytokines, antibodies or small molecules kinase inhibitors within 3 weeks or nitrosoureas/mitomycin C within 6 weeks] prior to allocation. Prior liver surgery or local treatment of metastases is allowed if there is an unequivocal progression.

   Note: Participants must have recovered from all AEs due to previous therapies to ≤Grade 1 or baseline. Participants with ≤Grade 2 neuropathy may be eligible.

   Note: Do not administer for at least 2 weeks following major surgery and until adequate wound healing.
4. Has received prior radiotherapy within 2 weeks of start of study intervention. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
5. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. Only mRNA vaccines are authorized to prevent SARS-CoV-2 infection (COVID-19) during the trial.
6. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
8. Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 2 years.

   Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, or other in-situ cancers
9. Has known active CNS metastases and/or carcinomatous meningitis. Brain imaging is not required at inclusion if asymptomatic. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention.
10. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or lenvatinib and/or any of their excipients.
11. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
12. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
13. Has an active infection requiring systemic therapy. Patients requiring systemic antibiotics for infection must have completed therapy at least 1 week prior to the first dose of study drug.
14. Has a known history of Human Immunodeficiency Virus (HIV) infection. HIV testing is not required at allocation.
15. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
16. Has a known history of active TB (Bacillus Tuberculosis).
17. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
18. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
19. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
20. Has had an allogenic tissue/solid organ transplant.
21. Concurrent or recent (less than 1 week prior inclusion) immunosuppressive medications (including corticosteroids exceeding 10 mg daily of prednisone equivalent, azathioprin); hydrocortisone at physiological doses is allowed;
22. Uncontrolled blood pressure (Systolic BP>150 mmHg and/or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication.
23. Electrolyte abnormalities that have not been corrected as assessed by the investigator.
24. Significant cardiovascular impairment: history of congestive heart failure from New York Heart Association (NYHA) Class III or IV, unstable angina, myocardial infarction or stroke within 12 months of the first dose of study drug, or cardiac arrhythmia with hemodynamic instability. Note : medically controlled arrhythmia would be permitted.
25. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy.
26. Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
27. Subjects who have not recovered adequately from any toxicity from other anti-cancer treatment regimens and/or complications from major surgery prior to starting therapy.
28. Has had major surgery within 3 weeks prior to first dose of study interventions. Note: Adequate wound healing after major surgery must be assessed clinically, independent of time elapsed for eligibility.
29. Has preexisting ≥Grade 3 gastrointestinal or non-gastrointestinal fistula
30. Has a LVEF below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO).
31. Prolongation of QTcF interval to >480 ms.
32. Gastrointestinal malabsorption or any other condition that might affect the absorption of lenvatinib
33. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-11-15 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) according to RECIST 1.1 criteria | After 9 cycles (i.e. 27 weeks +/- 2 weeks)
  PFS will be estimated as a crude rate at 27 weeks (+/- 2 weeks, i.e. 14 days) after the start of treatment. Will be considered progression events: objective clinical progression, radiological progression according to RECIST 1.1 criteria and death from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of first study treaments intakes until the date of first documented progression assessed up to 30 months
  PFS is defined as the time from the date of treatment start until the date of first objective clinical or radiological disease progression (RECIST 1.1) or death. Patients alive and without progression at the date of last contact will be censored at this date.
Objective response rate (ORR) | After 9 cycles (i.e. 27 weeks +/- 2 weeks)
  Objective response rate using the RECIST criteria version 1.1 is defined as a Confirmed complete response (CR) or partial response (PR) at nine cycles, 27 weeks (+/- 2 weeks, i.e. 14 days)
Progression-free survival (PFS) using the iRECIST criteria | After 9 cycles (i.e. 27 weeks +/- 2 weeks)
  27-weeks PFS using the iRECIST criteria, based on investigator assessment
Overall Survival (OS) | From date of first study treatments intake until the date of death from any cause, assessed up to 100 months
  OS is defined as the time from the date of treatment start until the date of death due to any cause. Patients alive at the date of last contact will be censored at this date.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rodrigues, MD, Principal Investigator — Institut Curie
Locations (1):
- Institut Curie, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).